CLINICAL TRIAL: NCT01305616
Title: Effect of Yellow-Tinted Intraocular Lens on Standard Automated Perimetry (SAP) and Short-wavelength Automated Perimetry (SWAP) in Patients With and Without Glaucoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rassoul Akram Hospital (Other)
Responsible Party: Naveed Nilforushan, Rassoul Akram Hospital,Ophthalmic Research Center,Department of Ophthalmology,Iran University of Medical Sciences
Allocation: Non-Randomized | Model: Parallel | Masking: None
Other Study IDs: 975
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2011-03-28 (Estimated); Status verified 2008-03

CONDITIONS: Cataract; Glaucoma
Keywords: Open angle Glaucoma; Yellow-tinted intraocular lens; Short-wavelength Automated Perimetry (SWAP); Standard Automated Perimetry (SAP); cataract
MeSH Terms: conditions — Cataract; Glaucoma; Glaucoma, Open-Angle | interventions — Phacoemulsification

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Group 1, glaucoma and cataract (Active Comparator): Group1 were those patients with visually significant cataract (less than grade 2) and mild to moderate open angle glaucoma
  Interventions: Procedure: Phacoemulsification with yellow-tinted intraocular lens
- Group2, cataract patients (Sham Comparator): This group included those patients with visually significant cataract and normal other eye examination.
  Interventions: Procedure: Phacoemulsification with yellow-tinted intraocular lens

INTERVENTIONS:
Procedure: Phacoemulsification with yellow-tinted intraocular lens — Phacoemulsification is a kind of cataract surgery using ultrasound machine. Yellow-tinted intraocular lens are a sort of lens with the ability to filter blue and ultraviolet spectrum of light (380-500 nanometer)
  Other Names: bluelight filteing intraocular lens
  Arms: Group 1, glaucoma and cataract
Procedure: Phacoemulsification with yellow-tinted intraocular lens — Phacoemulsification is a kind of cataract surgery using ultrasound machine. Yellow-tinted intraocular lens are a sort of lens with the ability to filter blue and ultraviolet spectrum of light.
  Other Names: bluelight filteing intraocular lens
  Arms: Group2, cataract patients

SUMMARY:
To investigate the effect of yellow-tinted IOLs on the Short Wave-length Automated Perimetry (SWAP) and Standard Automated Perimetry (SAP) in patients with and without glaucoma.

DETAILED DESCRIPTION:
Glaucoma is mostly a disease of old people and is highly accompanied with cataract.Some of these patients may need to perform cataract surgery during the course of glaucoma. But in glaucoma patients, the effect of cataract surgery and/or type of implanted intraocular lens (IOL) on the results of specific visual field tests, like SWAP, is still not well studied.From the past decade, various yellow-tinted IOLs with the speculation of protecting the retinal photoreceptors and decreasing the incidence of age-related macular degeneration have been introduced.These blue-light-filtering IOLs contain a yellow chromophore that filters ultra violet (UV) and a larger part of the high-energetic visible blue-light between 380 and 500 nm. Based on previous studies yellow-tinted IOLs decrease the amount of light transmission to the retina which may theoretically affect perimetry results. This might be even more important in patients with glaucoma where the sensitivity of test locations has decreased per se.

Since early diagnosis of glaucoma and its progression is highly dependent on visual field results, it is important to evaluate the effect of these IOLs on perimetry, particularly on SWAP, in which the blue-light-filtering IOLs might interfere with its findings.

ELIGIBILITY:
Inclusion Criteria:

* In group 1, visually significant cataract associated with well controlled mild to moderate open angle glaucoma (intraocular pressure < 18 with maximally-tolerated medical treatment)and no history of previous intraocular surgeries
* In group 2- Normal ophthalmic examination other than visually significant cataract

Exclusion Criteria:

* Diabetes mellitus
* neurological disease which may affect the results of visual field
* known systemic medication with involvement on visual field
* spherical refractive error less than -5 and more than +5 diopter
* cylindrical correction more than 3 diopter

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-05; Primary Completion 2009-11 (Actual); Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Mean deviation changes on SAP and SWAP before and after surgery | 2.5months
  Mean deviation(decibel) which is the average change of visual field points from normal age- matched group ,was obtained from visual field print out. Its value is from 0 to -30 decibels where the lower values means the point is more damaged.

SECONDARY OUTCOMES:
Visual Acuity changes measured with Snellen chart and Pattern Standard Deviation (PSD)and Foveal threshold (FT) changes on SAP and SWAP. | 2.5 months
  visual acuity measurements were converted to logarithm minimum angle of resolution (logMAR).PSD (decibel)and FT(decibel) were obtained from the Humphrey visual field machine printout.

CONTACTS AND LOCATIONS:
Overall Officials: Naveed Nilforushan, M.D, Principal Investigator — Rassoul Akram hospital,Department of Ophthalmology,Iran University of Medical Sciences
Locations (1):
- Rassoul Akram Hospital, Tehran, Tehran Province, Iran

REFERENCES:
- [Background] Jang SY, Ohn YH, Kim SW. Effect of yellow-tinted intraocular lenses on short-wavelength automated perimetry. Am J Ophthalmol. 2010 Aug;150(2):243-247.e1. doi: 10.1016/j.ajo.2010.02.023. PMID 20525530
- [Background] Kara-Junior N, Jardim JL, de Oliveira Leme E, Dall'Col M, Susanna R Jr. Effect of the AcrySof Natural intraocular lens on blue-yellow perimetry. J Cataract Refract Surg. 2006 Aug;32(8):1328-30. doi: 10.1016/j.jcrs.2006.03.033. PMID 16863969